CLINICAL TRIAL: NCT01711762
Title: A Phase 1 Study to Investigate the Absorption, Metabolism, and Excretion of [14C]-GDC-0973 Following Single Oral Dose Administration in Healthy Male Subjects
Brief Title: A Pharmacokinetics Study of Radioactive-Labeled GDC-0973 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: GP28369
Record Dates: First submitted 2012-10-18; First posted 2012-10-22 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — cobimetinib

ARMS (1):
- GDC-0973 Single Arm (Experimental)
  Interventions: Drug: GDC-0973

INTERVENTIONS:
Drug: GDC-0973 — Single oral dose of [14C]-GDC-0973

SUMMARY:
This open-label, non-randomized study will assess the absorption, metabolism, and excretion of radioactive-labeled [14C]-GDC-0973 in healthy male volunteers. Volunteers will receive a single dose of [14C]-GDC-0973.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5 and 29.9 kg/m2, inclusive
* No clinically significant findings from medical history, 12-lead ECG, and vital signs and laboratory evaluations
* Negative test for selected drugs of abuse
* No infection with hepatitis B, hepatitis C, human immunodeficiency virus (HIV)
* Sterile or agree to use an adequate contraception method
* Historically able to produce a minimum of 1 bowel movement per day

Exclusion Criteria:

* Significant history or clinical manifestation of any significant metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance unless approved by the Investigator
* History of stomach or intestinal surgery or resection (including a cholecystectomy) that would potentially alter absorption and/or excretion of orally administered drugs except that appendectomy and/or hernia repair will be allowed
* History of Gilbert's Syndrome
* History of diabetes mellitus and/or elevated fasting glucose at baseline
* History or presence of an abnormal ECG
* History of alcoholism or drug addiction within 1 year prior Check-in
* Participation in more than one other radiolabeled investigational study drug trial within 12 months prior to Check-in
* Exposure to significant radiation within 12 months prior to Check-in study drug occurred within 5 half-lives or 30 days, whichever is longer, prior to Check-in
* Use of any tobacco-containing or nicotine-containing products within 6 months prior to Check-in
* Participation in any other investigational study drug or biologic agent trial in which receipt of an investigational study drug occurred within 5 half-lives or 30 days, whichever is longer, prior to Check-in
* Use of any prescription medications/products within 14 days prior to Check-in

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2012-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Route of elimination of [14C]-GDC-0973 | approximately 8 weeks
Pharmacokinetics: maximum observed concentration (Cmax) | approximately 8 weeks
Pharmacokinetics: time to maximum concentration (tmax) | approximately 8 weeks
Pharmacokinetics: area under the concentration-time curve | approximately 8 weeks
Pharmacokinetics: apparent terminal elimination phase rate constant | approximately 8 weeks
Pharmacokinetics: apparent terminal elimination phase half-life | approximately 8 weeks
Pharmacokinetics: apparent total clearance | approximately 8 weeks
Pharmacokinetics: apparent volume of distribution | approximately 8 weeks
Pharmacokinetics: amount total radioactivity in whole blood/urine/feces | approximately 8 weeks

SECONDARY OUTCOMES:
Pharmacokinetics: quantification of GDC-0973-related metabolites in plasma, urine and fecal homogenates | approximately 8 weeks
Pharmacokinetics: plasma concentration of GDC-0973 | approximately 8 weeks
Safety: incidence of adverse events | approximately 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (1):
- Madison, Wisconsin, United States